CLINICAL TRIAL: NCT07034638
Title: Effects of White and Pink Noise Applied Before and During Colonoscopy on Pain and Anxiety: A Randomized Controlled Trial
Brief Title: Effects of White and Pink Noise Applied Before and During Colonoscopy on Pain and Anxiety
Acronym: Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Seda Cansu Yeniğün, Lecturer Dr, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Scy120991
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Surgical Procedures, Elective; Nurse Based Care Management
Keywords: colonoscopy; white noise; pink noise; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Patients in the control group will only be subject to the hospital's current standard care protocol. The procedures performed within the scope of this protocol include routine practices such as informing the patient, making the necessary medical preparations, and providing basic nursing interventions during the procedure. After the colonoscopy procedure is completed, the patient will be taken out of the endoscopy room and taken to the rest area where they will rest for 10 minutes in a quiet environment. At the end of this period, the VAS and VAS-A forms will be filled in again by the researcher and post-procedure pain and anxiety levels will be measured.
- white noise (Experimental): In this group, patients will listen to white noise via headphones in addition to the hospital's standard care protocol prior to and during the colonoscopy procedure, as directed by the researcher. White noise is a type of sound that contains equal intensity sound across the entire frequency spectrum and suppresses environmental sounds that distract the individual by masking external noise. Patients will choose one of three compact discs containing white noise (babbling brook, distant thunderstorm, soothing rain; Pure White Noise, Windsor, CO). The patient will listen to the noise via headphones for 20 minutes before the colonoscopy begins. It will continue uninterrupted throughout the procedure, and pain will be assessed with VAS and anxiety levels will be assessed with VAS-A during the procedure. The sound level will be adjusted to predetermined safe levels so as not to disrupt the patient's comfort. After the colonoscopy procedure is completed, the patient will be taken out of the e
  Interventions: Behavioral: WNG
- Pink noise (Experimental): In addition to the standard care protocol, the patients included in this group will listen to pink noise through headphones as directed by the researcher. Pink noise is a sound form that is dominated by low-frequency sounds and provides a more natural, soft acoustic environment. Sounds similar to sounds in nature (e.g. wind, rain, ocean waves) are included as pink noise. The patient will listen to pink noise through headphones for 20 minutes before the colonoscopy begins. It will continue uninterrupted throughout the procedure. During the procedure, pain will be assessed with VAS and anxiety levels will be assessed with VAS-A. The sound level will be adjusted to predetermined safe levels so as not to disrupt the patient's comfort. After the colonoscopy procedure is completed, the patient will be taken out of the endoscopy room and taken to the resting area where they will rest for 10 minutes in a quiet environment. At the end of this period, the researcher will fill in the VAS and VAS
  Interventions: Behavioral: PNG

INTERVENTIONS:
Behavioral: WNG — In addition to the hospital's standard care protocol, patients in this group will listen to white noise through headphones before and during the colonoscopy procedure, as directed by the researcher.
  Arms: white noise
Behavioral: PNG — In addition to the standard care protocol, patients included in this group will listen to pink noise through headphones as directed by the researcher.
  Arms: Pink noise

SUMMARY:
In recent years, there has been an increase in the use of endoscopic procedures due to the increase in diseases. Colonoscopy is widely used in the screening and diagnosis of many diseases, especially colorectal cancer. However, colonoscopy is perceived as an invasive, painful and uncomfortable procedure by patients. Moreover, it can cause pain associated with embarrassment, fear, anxiety and physical and emotional discomfort.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of white and pink noise applied before and during colonoscopy on pain and anxiety levels of patients. Colonoscopy is a widely used method in colon cancer screening and diagnosis and treatment of lower gastrointestinal system diseases; however, pain may occur in patients due to mesenteric distension and spasms during the procedure. In addition, many patients experience moderate anxiety during the procedure. Since pharmacological pain and anxiety management strategies may lead to some complications, in recent years, there has been an increase in the use of non-pharmacological methods such as music, video, virtual reality and distraction techniques. One of these methods, sound therapy, provides relaxation by directing the individual's attention to positive emotions. While white noise is a constant-intensity sound similar to the sound of the ocean or wind, pink noise resembles rain or rustling leaves with its lower frequency and soothing properties. There are a limited number of studies in the literature examining the effects of white and pink noise, but there is no study evaluating both types of noise together in colonoscopy patients. In order to fill this gap, the effects of white and pink noise on pain and anxiety are comparatively examined in this study.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,

  * Being over 18 years old,
  * Being able to speak and read and write Turkish,
  * The patient should not have a hearing problem,
  * Being conscious, oriented and cooperative

Exclusion Criteria:

* The patient's use of anxiolytics or analgesics on the day of the procedure,
* The patient's diagnosis of any psychiatric / neurological disease,
* The patient's preference for general anesthesia will be considered as exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2025-06-24 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Visual Anxiety Scale (VAS-A) | before colonoscopy 30 minutes
  VAS-A is a single-item measurement tool that has been used for psychological assessment since the beginning of the 20th century. It is frequently used in the assessment of pain, quality of life and mood. It was developed by "Cline et al" (1992) and is extremely simple, reproducible and requires minimal tools. The scale consists of a 10 cm long horizontal line with the labels "No anxiety" on the left and "I feel a lot of anxiety" on the right. The patient's anxiety level is calculated by measuring the distance between the leftmost part of the scale and the specified point. As the anxiety level approaches 10, anxiety increases.
Visual Anxiety Scale (VAS-A) | before colonoscopy 10 minutes
  VAS-A is a single-item measurement tool that has been used for psychological assessment since the beginning of the 20th century. It is frequently used in the assessment of pain, quality of life and mood. It was developed by "Cline et al" (1992) and is extremely simple, reproducible and requires minimal tools. The scale consists of a 10 cm long horizontal line with the labels "No anxiety" on the left and "I feel a lot of anxiety" on the right. The patient's anxiety level is calculated by measuring the distance between the leftmost part of the scale and the specified point. As the anxiety level approaches 10, anxiety increases.
The Visual Analog Scale (VAS) | before colonoscopy 30 minutes
  The Visual Analog Scale (VAS) is a single-dimensional scale commonly used to measure pain intensity. VAS is a measuring tool with a length of 0-10 cm (0-100 mm). This measuring tool can be used horizontally or vertically. The scale starts with "no pain" and ends with "unbearable pain". High scores obtained from the scale indicate high pain intensity. The cut-off points for pain scores obtained from the scale are recommended as 0-4 mm "no pain", 5-44 mm "mild pain", 45-74 mm "moderate pain" and 75-100 mm "severe pain".
The Visual Analog Scale (VAS) | before colonoscopy 10 minutes
  The Visual Analog Scale (VAS) is a single-dimensional scale commonly used to measure pain intensity. VAS is a measuring tool with a length of 0-10 cm (0-100 mm). This measuring tool can be used horizontally or vertically. The scale starts with "no pain" and ends with "unbearable pain". High scores obtained from the scale indicate high pain intensity. The cut-off points for pain scores obtained from the scale are recommended as 0-4 mm "no pain", 5-44 mm "mild pain", 45-74 mm "moderate pain" and 75-100 mm "severe pain".

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Cansu Yeniğün, Antalya, Kumluca, Turkey (Türkiye)